CLINICAL TRIAL: NCT06458075
Title: Intervention to Improve Patient-provider Communication and Medication Adherence Among Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Intervention to Improve Communication and Medication Adherence in Lupus
Acronym: CO-LEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00115358; 1R01MD018977-01 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control clinicians will continue usual care.
- CO-LEAD (Active Comparator): CO-LEAD clinicians will receive training in the intervention.
  Interventions: Behavioral: CO-LEAD

INTERVENTIONS:
Behavioral: CO-LEAD — The investigators will provide clinicians with a program to teach them to use effective communication strategies with patients to review real-time pharmacy refill data and the DOSE-Nonadherence-SLE survey, and engage and formulate solutions to adherence barriers together. The study team will provide the clinician intervention training in-person or virtually and will include didactics, demonstration, and practice that include two one-hour sessions one month apart. After training, CO-LEAD clinicians will be encouraged to incorporate the intervention in regular clinic visits with all patients.
  Arms: CO-LEAD

SUMMARY:
CO-LEAD is an intervention to improve patient-provider communication and medication adherence among patients with systemic lupus erythematosus (SLE).

The purpose of this study is to optimize the culturally appropriate delivery and test the effect of the CO-LEAD intervention, which includes the following:

1. clinicians will be provided with a program to teach them to use effective communication strategies with patients to review real-time pharmacy refill date, engage and formulate solutions to adherence barriers, and collaboratively overcome adherence barriers.
2. use of a reliable and valid patient-reported measure of the extent of and reasons for nonadherence that helps patients identify and communicate their adherence barriers with clinicians proactively, efficiently, and comprehensively.

DETAILED DESCRIPTION:
Substantial racial disparities exist in patients with systemic lupus erythematosus (SLE), a disease that markedly reduces life expectancy and quality of life. Long-term, consistent use of immune-altering medicines is critical for treating symptoms and preventing organ damage from SLE, but Black patients have lower medication adherence. While reasons for nonadherence are complex, Black patients with SLE are disproportionately affected by motivational barriers related to their beliefs, attitudes, and trust. Effective and collaborative patient-clinician communication can lead to more honest exchange of information, strengthen trust and therapeutic alliance, and thereby increase medication adherence and improve health outcomes. Unfortunately, effective patient-clinician discussions about nonadherence occur sporadically, and Black patients experience worse communication with their clinicians. Existing adherence interventions in SLE do not address patient-clinician communication nor focus on reducing racial disparities.

In this study, clinicians will go through training on how to assess medication adherence and communicate more effectively with this population. Clinicians will familiarize with EMR pharmacy refill data and the DOSE-Nonadherence-SLE questionnaire, a validated measure of the extent of and reasons for nonadherence. Clinicians will practice having a medication nonadherence discussion with another clinician in the intervention arm and give each other feedback after the practice. Clinicians will also be provided with resource handouts for medication adherence. The training will increase clinicians' confidence in conducting the intervention, and gain empathy role-playing as the patient. CO-LEAD team members will observe and give feedback to clinicians in real time.

The study will assess both communication and adherence outcomes.

ELIGIBILITY:
Clinician Inclusion Criteria:

1. Adult rheumatology attendings, advanced practice providers, and fellows at the two academic institutions
2. Clinicians who have ambulatory rheumatology care at least ½ day per week

Clinician Exclusion Criteria:

1. Clinicians at Duke University who were involved in the investigators' pilot work
2. Clinicians with an anticipated departure from the institution in the 12 months following enrollment

Patient Inclusion Criteria:

1. 18 years or older
2. English-speaking, able to provide consent
3. Diagnosed with SLE and receiving care with enrolled clinicians
4. Prescribed at least one SLE medication, and filling their SLE mediations at a pharmacy linked to Surescripts reporting visible in Epic EMR.

Patient Exclusion Criteria:

1. Non-English speakers
2. Patients who are prescribed only corticosteroids for SLE
3. Patients who are accompanied by third-party member that is not willing or able to remain in the waiting room during the patient's visit and

   * Does not wish to be audio recorded
   * A minor without a parental/legal guardian and/or
   * Unable to give consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of adherence discussions | During intervention period (up to 2 years)
  Proportion of SLE patient visits in which a nonjudgmental, patient-centered adherence discussion took place as determined by analysis of clinic visit audio recordings

SECONDARY OUTCOMES:
Quality of patient-clinician communication determined by audio recordings | During intervention period (up to 2 years)
  Audio recordings of clinic visits which will be analyzed using a validated coding scheme
Quality of patient-clinician communication determined by surveys | During intervention period (up to 2 years)
  The Interpersonal Processes of Care survey will be used
Change in SLE medication adherence | Baseline and post-intervention (up to 6 months)
  Determined by pharmacy refill data. Proportion of days covered (PDC) will be calculated as total days of supply dispensed.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Sun, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No